CLINICAL TRIAL: NCT04207372
Title: Determination of Protein Digestibility of Whey and Zein in Ileostomates
Brief Title: Protein Digestibility of Whey and Zein.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Massey University (Other); Global Dairy Platform Incorporated (Unknown)
Responsible Party: Principal Investigator, Geleijnse, Prof. Dr., Wageningen University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NL63446.081.17
Record Dates: First submitted 2019-11-28; First posted 2019-12-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Biological Availability
Keywords: Digestibility; Whey; Zein; Protein; Ileostomates
MeSH Terms: interventions — Zein

STUDY DESIGN:
Intervention Model Description: Intervention study with 6 test days, testing 3 meals each twice
Who Masked: Participant
Masking Description: Allocation of different proteins(or no protein) is blinded from participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whey protein isolate (Experimental)
  Interventions: Dietary Supplement: whey protein isolate
- Zein (Experimental)
  Interventions: Dietary Supplement: Zein
- Protein-free (Placebo Comparator)
  Interventions: Other: protein-free

INTERVENTIONS:
Dietary Supplement: whey protein isolate — whey protein isolate
  Arms: Whey protein isolate
Dietary Supplement: Zein — zein protein
  Arms: Zein
Other: protein-free — protein free
  Arms: Protein-free

SUMMARY:
The evaluation of protein quality has top priority according to Food and Agricultural Organization of the United Nations. However, one aspect of protein quality, namely the digestibility of protein is largely unknown. A database on this matter is lacking as it is difficult to measure ileal digestibility in humans.

DETAILED DESCRIPTION:
Objective: This study aims to determine the digestibility of amino acids in two protein sources in men and women with normally functioning ileostomies.

Study design: Intervention study with 6 test days, testing 3 meals each twice. Study population: Eight men and women with normally functioning ileostomies will be recruited for the study.

Intervention: On six separate test days, subjects will receive a meal, consisting of a drink and biscuit. With this, two different protein containing meals, i.e. zein and whey, and a protein-free meal is tested; these three treatments are given at two occasions, thus in total 6 meals are tested. After consumption of the meal, subjects collect their digesta for nine hours.

Main study parameters/endpoints: Ileal amino acid digestibility of zein and whey protein isolate.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The subject will not benefit from the study except for the contribution to scientific research. The risk of participating to this study is low, some gastrointestinal discomfort could occur. Subjects have to come to the research facility seven times, a screening visit of 1 hour, and 6 experimental days of 10 hours. Subjects will be financially compensated for participation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age between 18 and 60
* Willing to eat animal protein
* Have a well-established and normally functioning terminal ileostomy, with stomal faeces of normal physiological consistency
* Good general health, meaning subjects should be well-recovered from the ileostomy operation, their underlying disease should be cured or in remission and they should not have any other major health problems

Exclusion Criteria:

* Taken antibiotics or medication that majorly impair small intestinal digestion and absorption within eight weeks of participating in the study.
* Have been pregnant or breastfeeding in the last 12 months, or plan to become pregnant during the study
* Having renal impairment, coeliac disease or diabetes
* Drug abuse
* Alcohol consumption of >14 units per week.
* Having an allergy or intolerance to dairy, corn products or fructose
* Currently taking protein supplements and would not be willing to stop using these during the study
* Being on a controlled diet or dietary weight loss regimen during the two weeks prior to the start of this study and/or during the study
* Personnel of division of Human Nutrition, Wageningen University..
* Current participation in other research from the Division of Human Nutrition
* Not having a general practitioner

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
the ileal amino acid digestibility of Zein and Whey Protein Isolate | 9 hours per day
  ileal digesta samples are collected in the nine hours after consumption of these proteins and after consumption of a protein-free diet.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Human Nutrition, Wageningen University, Wageningen, Gelderland, Netherlands

REFERENCES:
- [Derived] van der Wielen N, de Vries S, Gerrits WJ, Lammers-Jannink K, Moughan PJ, Mensink M, Hendriks W. Presence of Unabsorbed Free Amino Acids at the End of the Small Intestine Indicates the Potential for an Increase in Amino Acid Uptake in Humans and Pigs. J Nutr. 2023 Mar;153(3):673-682. doi: 10.1016/j.tjnut.2023.01.038. Epub 2023 Feb 9. PMID 36809852